CLINICAL TRIAL: NCT02748629
Title: Randomized Controlled Single-Center Trial: Self-Gripping ProGrip Mesh Repair vs Lichtenstein Operation of Inguinal Hernia
Brief Title: ProGrip Mesh Repair vs Lichtenstein Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Health Center in Kartuzy, Poland (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKBNN/258/2015
Record Dates: First submitted 2016-04-12; First posted 2016-04-22 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; mesh; lichtenstein; hernia repair; selfgripping mesh
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ProGrip Mesh Repair (Active Comparator): 80 patients are randomized to inguinal hernia repair using selfgripping ProGrip Mesh (Covidien Parietex ProGrip Self-Fixating Mesh) - sutureless fixation.
  Interventions: Device: Covidien Parietex ProGrip Self-Fixating Mesh
- Lichtenstein Operation (Active Comparator): 80 patients are randomized to inguinal hernia repair using lightweight polypropylene mesh (<40 g/m2) with standard Lichtenstein technique.
  Interventions: Device: Lightweight Polypropylene Mesh (<38g/m2 after absorption)

INTERVENTIONS:
Device: Covidien Parietex ProGrip Self-Fixating Mesh
  Arms: ProGrip Mesh Repair
Device: Lightweight Polypropylene Mesh (<38g/m2 after absorption) — Serag Wiessner SERAMESH® PA 15x10 cm
  Arms: Lichtenstein Operation

SUMMARY:
The purpose of this trial is to compare clinical outcomes and to analyze cost-effectiveness following self-gripping, sutureless Parietex ProGrip Mesh to traditional Lichtenstein Operation with lightweight polypropylene mesh.

DETAILED DESCRIPTION:
Single-center patient-blinded randomized clinical trial comparing self-gripping mesh (Parietex ProGrip) and standard Lichtenstein method using lightweight polypropylene mesh. Patients will be randomly allocated to the Lichtenstein Operation (L) and ProGrip Repair (R) group. Patients will be followed for one year. The primary outcome measure are: postoperative pain using the Visual Analog Scale (VAS) and Numeric Rating Scale (NRS). Assessments will be made before the surgery, in the day of discharge, 1, 6 and 12 months postoperatively.

Secondary endpoints: recurrence rate, post-operative complications (short and long-term), foreign body sensation, incidence of surgical-site injury, costs, hospital stay, surgery duration, safety and patients satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary inguinal hernia
* Signed consent

Exclusion Criteria:

* Recurrent hernia
* Emergency procedure
* Patient not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative pain and its intensity using VAS Scale | 12 Months
  Assessment will be made using Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Rate of foreign body sensation - Subjective feeling of discomfort in the groin | 12 Months
  Foreign body sensation is a patients' subjective feeling of discomfort in the groin. Assesment will be made by phone questionnaire.
Hernia recurrence rate | 12 Months
  Recurrence rate is number of hernia recurrences after surgery (can only be diagnosed by surgeon via clinical examination)
Post-operative complications | 12 Months
  Short and Longterm complications: surgical site injury, hematoma, seroma, testicle ischemia, chronic pain)
Duration of surgery | Day of surgery
Incidence of Treatment-Emergent Adverse Events [Safety] | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz T Zamkowski, MD, Study Chair — Regional Health Center in Kartuzy, Department of General Surgery
Locations (1):
- Regional Health Center in Kartuzy, Kartuzy, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sanders DL, Nienhuijs S, Ziprin P, Miserez M, Gingell-Littlejohn M, Smeds S. Randomized clinical trial comparing self-gripping mesh with suture fixation of lightweight polypropylene mesh in open inguinal hernia repair. Br J Surg. 2014 Oct;101(11):1373-82; discussion 1382. doi: 10.1002/bjs.9598. Epub 2014 Aug 21. PMID 25146918